CLINICAL TRIAL: NCT04124393
Title: Comparing Right Colon Adenoma and Hyperplastic Polyp Miss Rates in Colonoscopy Using Water Exchange and CO2 Insufflation: A Multicenter Randomized Tandem Study
Brief Title: Multicenter Evaluation of Right Colon Polyp Miss Rates Using Water Exchange Versus CO2 Insufflation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evergreen General Hospital, Taiwan (Other)
Collaborators: Taipei Medical University Hospital (Other); Dalin Tzu Chi General Hospital (Other); Sepulveda Ambulatory Care Center, VA Greater Los Angeles Healthcare System (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EGH-2020
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Right Colon Adenoma Miss Rate; Right Colon Hyperplastic Polyp Miss Rate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The second endoscopist will perform tandem right colon examination and is blinded to the insertion method used by the first endoscopist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water Exchange (WE) Colonoscopy (Active Comparator): In the WE group, the air pump will be turned off before starting the procedure. During the insertion phase, the colon will be irrigated with warm water (32C-35C). WE entails the infusion of water to open the lumen and simultaneous suction if the endoscope has two channels, and sequentially if the endoscope has only one channel. When the cecum is reached and after most of the water is suctioned to collapse the cecal lumen, CO2 will be opened. The colonoscope will be withdrawn to the hepatic flexure. All polyps identified will be resected (colon polypectomy). The colonoscope will then be reinserted into the cecum by the first endoscopist. A tandem inspection of the right colon will be performed by a blinded endoscopist. All polyps found herein will be counted as the missed polyps. After the second withdrawal to the distal hepatic flexure, the remainder of the colon will be examined in a standard manner by the first endoscopist.
  Interventions: Procedure: Colon Polypectomy
- CO2 Insufflation Colonoscopy (Active Comparator): In the CO2 group, colonoscopy is performed in the usual fashion, with minimal insufflation required to aid insertion. Cleaning in the CO2 group will be performed entirely during withdrawal. Upon arriving at the cecum, CO2 insufflation will be used and the colonoscope will be withdrawn from the cecum to the hepatic flexure. All polyps identified will be resected (colon polypectomy). Then, the colonoscope will be reinserted into the cecum by the first endoscopist. A tandem inspection of the right colon will be performed by a blinded endoscopist. All polyps found herein will be counted as the missed polyps. After the second withdrawal to the distal hepatic flexure, the remainder of the colon will be examined in a standard manner by the first endoscopist.
  Interventions: Procedure: Colon Polypectomy

INTERVENTIONS:
Procedure: Colon Polypectomy — Polyp search and resection will be performed entirely during the withdrawal phase in both WE and CO2 groups. Insertion inspection and polypectomy will not be performed. All polyps in the proximal colon, defined as cecum, ascending colon, hepatic flexure, and transverse colon, will be removed irrespective of their size and appearance.

SUMMARY:
A prospective multicenter randomized controlled trial (RCT) comparing water exchange (WE) colonoscopy and carbon dioxide (CO2) insufflation in terms of right colon combined adenoma miss rate (AMR) and hyperplastic polyp miss rate (HPMR) by tandem inspection.

DETAILED DESCRIPTION:
This will be a prospective RCT comparing CO2 insufflation and WE in terms of right colon combined AMR and HPMR by tandem inspection. It will be a multicenter study conducted in three community hospitals (Evergreen General Hospital, Taoyuan; Dalin Tzu-Chi Hospital, Chiayi; Taipei Medical University Hospital, Taipei) in Taiwan. Consecutive patients aged 45 years or older undergoing colonoscopy for screening, surveillance, and positive FIT will be considered for enrollment from December 2019 to May 2021. A written informed consent will be obtained from all participating patients. Participants will be randomized in a 1:1 ratio to undergo either the CO2 insufflation colonoscopy (CO2 group) or WE colonoscopy (WE group). WE colonoscopies will be performed by five board-certified colonoscopists (Chi-Liang Cheng, Yen-Lin Kuo [Evergreen General Hospital]; Yu-Hsi Hsieh, Chih-Wei Tseng [Dalin Tzu-Chi Hospital]; Jui-Hsiang Tang [Taipei Medical University Hospital]. Standard colonoscopes (CF-Q260AL/I, CF-HQ290L/I; Olympus Medical Systems Corp., Tokyo, Japan) will be used. Felix W. Leung will be involved in the study design, data analyses, and report preparation, but not in patient enrollment. Antispasmodic medication will not be administered during colonoscopy examination. CO2 insufflation will be used for CO2 group and the withdrawal phase of the WE group. In the WE group, the air pump will be turned off before starting the procedure. During the insertion phase, air and residual water or feces in the rectum will be aspirated, and then the colon will be irrigated with warm water. When the cecum is reached and after most of the water is suctioned to collapse the cecal lumen, CO2 will be opened. In the CO2 group, colonoscopy is performed in the usual fashion, with minimal insufflation required to aid insertion. Cleaning in the CO2 group will be performed entirely during withdrawal. Upon arriving at the cecum, CO2 insufflation will be used in both groups and the scope will be withdrawn from the cecum to the hepatic flexure, with inspection of the mucosa at the same time. All polyps identified will be resected and sent for pathology evaluation. The most distal part of the hepatic flexure will be marked by a forceps biopsy and then the scope will be reinserted into the cecum by the first endoscopist using CO2 insufflation. A tandem inspection of the right colon will then be performed by a blinded endoscopist in both study groups. All polyps found herein will be counted as the missed polyps. After the second withdrawal to the mark of distal hepatic flexure, the remainder of the colon will be examined in a standard manner by the first endoscopist. Polyp search and resection will be performed during the withdrawal phase in both groups. Insertion polypectomy will not be performed.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients aged 45 years or older undergoing colonoscopy for screening, surveillance, and positive fecal immunochemical test will be considered for enrollment.

Exclusion Criteria:

* Familial adenomatous polyposis and hereditary non-polyposis colorectal cancer (CRC) syndrome, personal history of CRC or inflammatory bowel disease, previous colonic resection, obstructive lesions of the colon, gastrointestinal bleeding, allergy to fentanyl, midazolam or propofol, American Society of Anesthesiology classification of physical status grade 3 or higher, mental retardation, pregnancy, and refusal to provide a written informed consent.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Right Colon Adenoma Miss Rate | One day
  Lesions detected on the tandem right colon examination will be used for the calculation of adenoma miss rate. Right colon adenooma miss rate will be calculated as the the number of adenomas missed during the first right colon examination divided by the total number of adenomas detected during both the first and tandem right colon examinations.
Right Colon Hyperplastic Polyp Miss Rate | One day
  Lesions detected on the tandem right colon examination will be used for the calculation of hyperplastic polyp miss rate. Right colon hyperplastic polyp miss rate will be calculated as the the number of hyperplastic polyps missed during the first right colon examination divided by the total number of hyperplalstic polyps detected during both the first and tandem right colon examinations.

CONTACTS AND LOCATIONS:
Overall Officials: Chiliang Cheng, M.D., Principal Investigator — Evergreen General Hospital
Locations (1):
- Evergreen General Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] le Clercq CM, Bouwens MW, Rondagh EJ, Bakker CM, Keulen ET, de Ridder RJ, Winkens B, Masclee AA, Sanduleanu S. Postcolonoscopy colorectal cancers are preventable: a population-based study. Gut. 2014 Jun;63(6):957-63. doi: 10.1136/gutjnl-2013-304880. Epub 2013 Jun 6. PMID 23744612
- [Background] Fuccio L, Frazzoni L, Hassan C, La Marca M, Paci V, Smania V, De Bortoli N, Bazzoli F, Repici A, Rex D, Cadoni S. Water exchange colonoscopy increases adenoma detection rate: a systematic review with network meta-analysis of randomized controlled studies. Gastrointest Endosc. 2018 Oct;88(4):589-597.e11. doi: 10.1016/j.gie.2018.06.028. Epub 2018 Jul 5. PMID 29981753
- [Background] Leung FW, Koo M, Cadoni S, Falt P, Hsieh YH, Amato A, Erriu M, Fojtik P, Gallittu P, Hu CT, Leung JW, Liggi M, Paggi S, Radaelli F, Rondonotti E, Smajstrla V, Tseng CW, Urban O. Water Exchange Produces Significantly Higher Adenoma Detection Rate Than Water Immersion: Pooled Data From 2 Multisite Randomized Controlled Trials. J Clin Gastroenterol. 2019 Mar;53(3):204-209. doi: 10.1097/MCG.0000000000001012. PMID 29505552
- [Background] Cheng CL, Kuo YL, Hsieh YH, Tang JH, Leung FW. Water exchange colonoscopy decreased adenoma miss rates compared with literature data and local data with CO2 insufflation: an observational study. BMC Gastroenterol. 2019 Aug 14;19(1):143. doi: 10.1186/s12876-019-1065-2. PMID 31412789
- [Background] Zhao S, Wang S, Pan P, Xia T, Chang X, Yang X, Guo L, Meng Q, Yang F, Qian W, Xu Z, Wang Y, Wang Z, Gu L, Wang R, Jia F, Yao J, Li Z, Bai Y. Magnitude, Risk Factors, and Factors Associated With Adenoma Miss Rate of Tandem Colonoscopy: A Systematic Review and Meta-analysis. Gastroenterology. 2019 May;156(6):1661-1674.e11. doi: 10.1053/j.gastro.2019.01.260. Epub 2019 Feb 6. PMID 30738046
- [Derived] Cheng CL, Tang JH, Hsieh YH, Kuo YL, Fang KC, Tseng CW, Su IC, Chang CC, Tsui YN, Lee BP, Zou KY, Lee YS, Leung FW. Comparing Right-Sided Colon Adenoma and Serrated Polyp Miss Rates With Water Exchange and CO 2 Insufflation: A Randomized Controlled Trial. Am J Gastroenterol. 2024 Oct 30;120(7):1615-1623. doi: 10.14309/ajg.0000000000003168. PMID 39471473